CLINICAL TRIAL: NCT01256476
Title: A RANDOMIZED, DOUBLE-BLIND, ACTIVE CONTROLLED, PARALLEL GROUP STUDY OF PITAVASTATIN 4 MG VS. PRAVASTATIN 40 MG IN PATIENTS WITH PRIMARY HYPERLIPIDEMIA OR MIXED DYSLIPIDEMIA
Brief Title: Prevail-Us: A Study Of Pitavastatin 4 mg Vs. Pravastatin 40 mg In Patients With Primary Hyperlipidemia Or Mixed Dyslipidemia
Acronym: PREVAIL-US
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NK-104-4.04US
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2012-04-30 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Primary Dyslipidemia; Mixed Dyslipidemia
MeSH Terms: interventions — pitavastatin; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pitavastatin 4 mg once daily (QD) (Experimental)
  Interventions: Drug: pitavastatin
- pravastatin 40 mg once daily (QD) (Active Comparator)
  Interventions: Drug: pravastatin

INTERVENTIONS:
Drug: pitavastatin — pitavastatin 4 mg once daily (QD)
  Other Names: Livalo
  Arms: pitavastatin 4 mg once daily (QD)
Drug: pravastatin — Pravastatin 40 mg once daily (QD)
  Arms: pravastatin 40 mg once daily (QD)

SUMMARY:
Randomized, double-blind, double-dummy, 12-week, active-controlled study of pitavastatin 4 mg daily(QD) vs. pravastatin 40 mg daily(QD) in subjects with primary hyperlipidemia or mixed dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with primary hypercholesterolemia or mixed dyslipidemia who are ≥18 and ≤80 years of age at the time of consent
* Plasma Low-density lipoprotein cholesterol (LDL-C) ≥130 milligrams per deciliter (mg/dL) and ≤220 mg/dL and triglyceride (TG) levels of ≤400 mg/dL

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* Any conditions which may cause secondary dyslipidemia
* Uncontrolled diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Huntsville, Alabama
  - Muscle Shoals, Alabama
  - Chandler, Arizona
  - Goodyear, Arizona
  - Phoenix, Arizona
  - Beverly Hills, California
  - Los Angeles, California
  - Newport Beach, California
  - Colorado Springs, Colorado
  - Clearwater, Florida
  - DeLand, Florida
  - Fort Luaderdale, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Oviedo, Florida
  - Pembroke Pines, Florida
  - Ponte Vedra, Florida
  - Addison, Illinois
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Erlanger, Kentucky
  - Baltimore, Maryland
  - Brockton, Massachusetts
  - Edina, Minnesota
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Rochester, New York
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Lyndhurst, Ohio
  - Willoughby Hills, Ohio
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Corpus Christi, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Olympia, Washington

REFERENCES:
- [Derived] Miller PE, Martin SS, Joshi PH, Jones SR, Massaro JM, D'Agostino RB, Sponseller CA, Toth PP. Pitavastatin 4 mg Provides Significantly Greater Reduction in Remnant Lipoprotein Cholesterol Compared With Pravastatin 40 mg: Results from the Short-term Phase IV PREVAIL US Trial in Patients With Primary Hyperlipidemia or Mixed Dyslipidemia. Clin Ther. 2016 Mar;38(3):603-9. doi: 10.1016/j.clinthera.2016.02.001. Epub 2016 Feb 26. PMID 26922296
- [Derived] Sponseller CA, Morgan RE, Kryzhanovski VA, Campbell SE, Davidson MH. Comparison of the lipid-lowering effects of pitavastatin 4 mg versus pravastatin 40 mg in adults with primary hyperlipidemia or mixed (combined) dyslipidemia: a Phase IV, prospective, US, multicenter, randomized, double-blind, superiority trial. Clin Ther. 2014 Aug 1;36(8):1211-22. doi: 10.1016/j.clinthera.2014.06.009. Epub 2014 Jul 3. PMID 24998014
- [Derived] Chapman MJ, Orsoni A, Robillard P, Hounslow N, Sponseller CA, Giral P. Effect of high-dose pitavastatin on glucose homeostasis in patients at elevated risk of new-onset diabetes: insights from the CAPITAIN and PREVAIL-US studies. Curr Med Res Opin. 2014 May;30(5):775-84. doi: 10.1185/03007995.2013.874989. Epub 2014 Jan 10. PMID 24328357

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pitavastatin 4 mg Once a Day (QD) | Pravastatin 40 mg Once a Day (QD)
Started | 164 | 164
Completed | 158 | 157
Not Completed | 6 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Persistent ALT or AST elevation | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Subject non-compliance | 0 | 1
Not completed — LDL-C elevation exceeding 250 mg/dL | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 4 mg Once a Day (QD) | Pravastatin 40 mg Once a Day (QD) | Total
Number analyzed (Participants) | 164 | 164 | 328
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 127 | 249
  >=65 years | 42 | 37 | 79
Age Continuous [Mean (Standard Deviation); unit: years] | 58.8 (8.93) | 57.0 (10.23) | 57.9 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 79 | 162
  Male | 81 | 85 | 166
Region of Enrollment [Number; unit: participants]
  United States | 164 | 164 | 328

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Low Density Lipoprotein Cholesterol(LDL-C) From Baseline to Week 12
Time Frame: Baseline and 12 weeks
Population: All randomized subjects who took at least 1 dose of double-blind study drug, had a baseline efficacy measurement, and had at least 1 valid post-baseline efficacy measurement.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Pitavastatin 4 mg Once Daily (QD) | Pravastatin 40 mg Once Daily (QD)
Number analyzed (Participants) | 161 | 161
percent | -34.8 (1.20) | -22.7 (1.22)

ADVERSE EVENTS:
Arm/Group | Pitavastatin 4 mg Once a Day (QD) | Pravastatin 40 mg Once a Day (QD)
Serious Adverse Events (participants affected / at risk) | 2/164 | 1/164
Other Adverse Events (participants affected / at risk) | 19/164 | 14/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg Once a Day (QD) (N=164) | Pravastatin 40 mg Once a Day (QD) (N=164)
appendicitis perforated (Gastrointestinal disorders) | 1 | 0
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg Once a Day (QD) (N=164) | Pravastatin 40 mg Once a Day (QD) (N=164)
upper respiratory tract infection (Infections and infestations) | 8 | 9
Nasopharyngitis (Infections and infestations) | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
May not publish.